CLINICAL TRIAL: NCT07343167
Title: Factors Associated With Mortality in Streptococcal Anginosus Bacteremia
Acronym: SGA
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9821
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Streptococcal Infections
Keywords: Streptococcal Infections; Streptococcal Anginosus Bacteremia; Streptococcal anginosus infections
MeSH Terms: conditions — Streptococcal Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Streptococcal anginosus infections (S. constellatus, S. anginosus, and S. intermedius) are characterized by their severity, linked to high mortality and frequent infectious complications. Several studies in the literature highlight this severity, with mortality rates estimated at around 15%.

The aim of this research is to identify the factors associated with mortality in Streptococcal anginosus bacteremia.

ELIGIBILITY:
Inclusion Criteria:

* Major subject (≥18 years old)
* Hospitalized between January 1, 2019, and December 31, 2024, in one of the participating centers
* Having presented during the study period at least one positive blood culture for Streptococcus anginosus, Streptococcus constellatus, or Streptococcus intermedius in a laboratory at a participating center

Exclusion Criteria:

* Refusal to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Major subject having presented during the study period at least one positive blood culture for Streptococcus anginosus, Streptococcus constellatus, or Streptococcus intermedius in a laboratory at a participating center
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03-08 (Estimated)

PRIMARY OUTCOMES:
28-day in-hospital mortality | 28-Day Mortality Following Streptococcal Infection
  28-Day In-Hospital Mortality Following Streptococcal Infection

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de référence des maladies vectorielles à tiques, CNR Borrelia - CHU de Strasbourg - France, Strasbourg, France